CLINICAL TRIAL: NCT01245400
Title: A Prospective, Randomized, Double-Blind, Multicenter Clinical Trial to Evaluate the Safety and Efficacy of the Z-Lig Medical Device Compared to Allograft for the Reconstruction of Ruptured Anterior Cruciate Ligaments
Brief Title: Safety and Efficacy Study of the Z-Lig Medical Device Compared to Allograft
Acronym: Z-Lig
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aperion Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABI-ZLig-01-10-01
Record Dates: First submitted 2010-11-01; First posted 2010-11-22 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Ruptured Anterior Cruciate Ligaments
Keywords: Z-Lig; allograft; ACL; Anterior Cruciate Ligament; ACLR; Anterior Cruciate Ligament Reconstruction; EU; European Union; S. Africa; Reconstruction of ruptured anterior cruciate ligaments
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Z-Lig (Experimental): Z-Lig Anterior Cruciate Ligament Reconstruction (ACLR) graft implantation performed under anesthesia during an arthroscopic procedure.
  Interventions: Device: Z-Lig
- Allograft (Active Comparator): Allograft bone/tendon graft implantation performed under anesthesia during an arthroscopic procedure.
  Interventions: Device: allograft

INTERVENTIONS:
Device: Z-Lig — ACL replacement
  Arms: Z-Lig
Device: allograft — ACL replacement
  Arms: Allograft

SUMMARY:
The purpose of this Trial is to demonstrate the safety and efficacy of the Investigational Device for the treatment of ruptured Anterior Cruciate Ligament (ACL) of the knee compared to Allograft.

DETAILED DESCRIPTION:
Current techniques to reconstruct ruptured ACLs utilize either autologous tissue or allograft (cadaver) tissue. Both treatments have well-documented shortcomings (i.e., autologous tissue exposes patients to increased morbidity and allograft tissue use is limited by global availability and quality).

There are currently no effective artificial materials or xenograft tissue substitutes widely available. The purpose of this multicenter clinical trial is to evaluate the safety and efficacy of the Z-Lig in Subjects who require reconstruction of primary ruptured anterior cruciate ligaments and compare those results to allograft.

ELIGIBILITY:
Contact Sponsor

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
KT-1000 | baseline, 3,6, 12 & 24 monhts
  Contact Sponsor

CONTACTS AND LOCATIONS:
Locations (6):
- Contact Sponsor, Belgium
- Contact Sponsor, Denmark
- Bologna, Italy
- Contact Sponsor, Netherlands
- Contact Sponsor, South Africa
- Contact Sponsor, Spain

REFERENCES:
- See also: Click here for more information about this study: Z-Lig compared to Allograft — http://www.aperionbiologics.com/